CLINICAL TRIAL: NCT06281405
Title: A Prospective Randomized Phase II Trial of CAPOX and PD-1 Antibody Combined With or Without Radiotherapy for Microsatellite Stable Locally Advanced Rectal Cancer (TORCH-iTNT)
Brief Title: CAPOX and PD-1 Antibody Combined With or Without Radiotherapy for MSS Locally Advanced Rectal Cancer
Acronym: TORCH-iTNT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Study Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2023-290-3409
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Rectal Cancer; Neoadjuvant Therapy
MeSH Terms: interventions — spartalizumab; toripalimab; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunochemotherapy group (Experimental): The patients will receive 6 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT while a W&W option can be applied to patients achieving cCR.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine
- Radiation plus immunochemotherapy group (Experimental): The patients will receive short-course radiotherapy (25Gy/5Fx), followed by 6 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT while a W&W option can be applied to patients achieving cCR.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Radiation: Short-course radiotherapy

INTERVENTIONS:
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg d1 q3w
  Other Names: Toripalimab
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid d1-14 q3w
Radiation: Short-course radiotherapy — Short-course radiotherapy: 25Gy/5Fx
  Arms: Radiation plus immunochemotherapy group

SUMMARY:
TORCH-iTNT is a prospective, multicentre, randomized phase II trial. 198 LARC (T3-4/N+M0, distance from anal verge ≤12cm) patients will be treated with total neoadjuvant therapy (TNT) and assigned to Group A and Group B (1:1). Group A receives 6 cycles of Toripalimab combined with CAPOX (ToriCAPOX). Group B receives SCRT (25Gy/5Fx) followed by 6 cycles of ToriCAPOX. TME surgery is scheduled after TNT while a watch and wait (W&W) option can be applied to patients achieving clinical complete response (cCR). The primary endpoint is complete response (CR, pathological complete response [pCR] plus cCR) rate. The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, organ or anal preservation rate, 3-year DFS rate, etc.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-70 years old, female and male;
2. Pathological confirmed adenocarcinoma;
3. The distance from anal verge ≤ 10 cm;
4. MSI/MMR status: MSS/pMMR;
5. Clinical stage T3-4 and/or N+, without distance metastases;
6. At least one of the following factors is present: distance from the anus ≤5 cm, cT4, cN2, positive cMRF, positive cEMVI, or positive lateral lymph nodes;
7. KPS ≥ 70;
8. No radiotherapy, chemotherapy, immunotherapy, or any other anti-tumor therapy had been administered prior to enrollment;
9. Baseline blood and biochemical indicators meet the following criteria: neutrophils ≥ 1.5 × 10^9/L, Hb ≥ 90 g/L, PLT ≥ 100 × 10^9/L, ALT/ AST ≤ 2.5 ULN, Cr ≤ 1 ULN;
10. With good compliance and signed the consent form.

Exclusion Criteria

1. Pregnancy or breast-feeding women;
2. Known history of other malignancies within 5 years;
3. Known history of severe neurological or mental illness (such as schizophrenia, dementia or epilepsy);
4. Current severe cardiac disease (cardiac dysfunction and arrhythmia), renal dysfunction and liver dysfunction;
5. Acute cardiac infarction or cerebral ischemic stroke occurred within 6 months before recruitment;
6. Uncontrolled infection which needs systemic therapy;
7. Active autoimmune disease or immunodeficiencies, known history of organ transplantation or systematic use of immunosuppressive agents;
8. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1 to 2 antibody positive), active syphilis infection, active pulmonary tuberculosis infection;
9. Allergic to any component of the therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 1 month after the surgery or the decision of W&W
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of cCR with W&W strategy.

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until 3 months after the completion neoadjuvant therapy
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
3 year organ or anal preservation rate | From date of randomization until the resection of rectum or anus, assessed up to 36 months.
  3 year organ or anal preservation rate
3 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3 year local recurrence free survival rate | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival
3 year distant metastasis free survival rate | From date of randomization until the date of first documented distant metastasis, assessed up to 36 months.
  Rate of 3 year distant metastasis free survival
3 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
Rate of surgical complications | The surgical complications were assessed within 3 months after the surgery.
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China